CLINICAL TRIAL: NCT01410162
Title: A Randomized, Open Label, Cross Over Study to Examine the Impact of Prograf and Advagraf on Tacrolimus Exposure, Mycophenolic Acid Pharmacokinetics, Renal Allograft Function or Adverse Effects.
Brief Title: Advagraf/Prograf Conversion Trial
Acronym: SG#153
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Norman Muirhead (Other)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Norman Muirhead, Professor, Medicine University of Western Ontario, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R-10-647; 17393 (Other: REB)
Record Dates: First submitted 2011-06-29; First posted 2011-08-04 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Renal Transplant; Kidney Pancreas Transplant
Keywords: Renal; Kidney/Pancreas; Transplant; conversion; bioequivalence; Mycophenolate Acid
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advagraf (Active Comparator)
  Interventions: Drug: Tacrolimus
- Prograf (Active Comparator)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — tacrolimus extended release capsules vs Prograf

SUMMARY:
Renal and kidney pancreas transplant patients will be randomized to once daily Advagraf or twice daily Prograf to assess changes in tacrolimus and mycophenolate mofetil exposure, renal allograft function, other relevant biochemical parameters and treatment related adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant or Renal Pancreas patients who are > 12 months post transplant
* Stable allograft function defined as eGFR > 30-60ml/min
* Renal patients who have a stable tacrolimus trough level of 5-8ng/ml in prior 3 months; Renal pancreas patients who have a stable tacrolimus trough level of 3-10 mg/ml in prior 3 months
* Receiving concomitant therapy with mycophenolate mofetil in a dose of 500-1000mg bid or equivalent

Exclusion Criteria:

* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
* History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
* Treated rejection within 3 months of randomization.
* Increased serum creatinine > 20% within 3 months of randomization.
* Subject is pregnant or breastfeeding
* Subject has significant co-morbid disease (eg. Malignancy or uncontrolled infection) or disability (e.g. cognitive deficit) which prevents understanding of, or adherence to, the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-12; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
renal function | baseline to 6 months

SECONDARY OUTCOMES:
Bioequivalence of MPA exposure with Advagraf | Baseline, 12 weeks and 24 weeks
  Bioequivalence is measured using Pharmacokinetic monitoring of MPA plasma concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Muirhead, Principal Investigator — London Health Sciences Centre Inc
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada